CLINICAL TRIAL: NCT01426373
Title: Multicenter, Open-label Study of ATX-101 (Sodium Deoxycholate Injection) for the Reduction of Localized Subcutaneous Fat in the Submental Area
Brief Title: Open-Label Study of Deoxycholic Acid for the Reduction of Localized Subcutaneous Fat in the Submental Area
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATX-101-11-26
Record Dates: First submitted 2011-08-26; First posted 2011-08-31 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Moderate or Severe Submental Fullness
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Deoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deoxycholic Acid 2 mg/cm² (Experimental): Participants received deoxycholic acid 2 mg/cm² administered in 0.2 mL injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
  Interventions: Drug: Deoxycholic acid injection

INTERVENTIONS:
Drug: Deoxycholic acid injection — Formulated as an injectable solution containing deoxycholic acid at a concentration of 10 mg/mL.
  Other Names: ATX-101; Kybella

SUMMARY:
To evaluate the safety of deoxycholic acid subcutaneous injections in the submental area (below the chin).

ELIGIBILITY:
Inclusion Criteria:

* Submental fat graded by the investigator as 2, 3, or 4 using the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) and graded by the subject as 2, 3, or 4 using the Patient-Reported Submental Fat Rating Scale (PR-SMFRS) as determined on visit 1 (within 28 days before the subject's first dosing session)
* Dissatisfaction with the submental area rated by the subject as 0, 1, or 2 using the Subject Self-rating Scale (SSRS) as determined on visit 1 (within 28 days before the subject's first dosing session)
* Males and nonpregnant, nonlactating females 18 years of age or greater, on the day of the subject's first dosing session (visit 2). Females of childbearing potential must have a negative human chorionic gonadotropin (serum) test result within 28 days before visit 2 and agree to practice adequate contraception, in the judgment of the investigator, during the course of the study
* A normal result on coagulation tests (prothrombin time (PT), partial thromboplastin time (PTT)) obtained within 28 days before subject's first dosing session
* History of stable body weight, in the judgment of the investigator, for at least 6 months before subject's first dosing session
* Expected to understand and comply with the visit schedule and all protocol-specified tests and procedures and agreement by the subject to refrain from making significant changes, in the judgment of the investigator, to his or her dietary or exercise habits during the course of the subject's participation
* Medically able to undergo the administration of study drug determined by clinical and laboratory tests obtained within 28 days before subject's first dosing session for which the investigator identifies no clinically significant abnormality
* Signed informed consent obtained before any study-specific procedure is performed

Exclusion Criteria:

* History of any intervention to treat submental fat (eg, liposuction, surgery, or lipolytic agents)
* History of trauma associated with the chin or neck areas, which in the judgment of the investigator may affect evaluation of safety or efficacy of treatment
* A grade of 4 on the Submental Skin Laxity Grading scale (SMSLG) or any other anatomical feature (eg, predominant subplatysmal fat, loose skin in the neck or chin area, prominent platysmal bands) for which reduction in submental fat may, in the judgment of the investigator, result in an aesthetically unacceptable outcome
* Evidence of any cause of enlargement in the submental area (eg, thyroid enlargement, cervical adenopathy) other than localized submental fat
* Body mass index of ≥ 40 kg/m² as determined on visit 1 (week 0)
* History or current symptoms of dysphagia
* Any medical condition that would interfere with assessment of safety or efficacy or compromise the subject's ability to undergo study procedures or give informed consent
* Treatment with radio frequency, laser procedures, chemical peels, or dermal fillers in the neck or chin area within 12 months before the first treatment session, or botulinum toxin injections in the neck or chin area within 6 months before the first treatment session
* History of sensitivity to any components of the study drug or to topical or local anesthetics (eg, lidocaine, benzocaine, novocaine)
* Previous treatment in this study or previous participation in a Kythera-sponsored ATX-101 study
* Treatment with an investigational device or agent within 30 days before the subject's first treatment session

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Beddingfield, III, M.D., PhD, Study Director — Kythera Biopharmaceuticals, Inc
Locations (18):
- United States (18):
  - Mark Rubin, Beverly Hills, California
  - Mitchel Goldman, La Jolla, California
  - Jeffrey Klein, San Juan Capistrano, California
  - Ava Shamban, Santa Monica, California
  - Steven Teitelbaum, Santa Monica, California
  - Susan Weinkle, Bradenton, Florida
  - Palm Beach Cosmetic, West Palm Beach, Florida
  - Steven Dayan, Chicago, Illinois
  - Lupo Center for Aesthetic and General Dermatology, New Orleans, Louisiana
  - Grekin Skin Institute, Warren, Michigan
  - David Goldberg, MD, Hillsborough, New Jersey
  - Roy Geronemus, MD, New York, New York
  - Macrene Alexiades-Armenakas, New York, New York
  - Sue Ellen Cox, Chapel Hill, North Carolina
  - Richard Fried, Yardley, Pennsylvania
  - Michael Gold, Nashville, Tennessee
  - Suzanne Bruce, Houston, Texas
  - Jeffrey Adelglass, Plano, Texas

REFERENCES:
- [Derived] Beer K, Weinkle SH, Cox SE, Rubin MG, Shamban A, Somogyif C. ATX-101 (Deoxycholic Acid Injection) for Reduction of Submental Fat: Results From a 12-Month Open-Label Study. J Drugs Dermatol. 2019 Sep 1;18(9):870-877. PMID 31524342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 18 investigational centers in the United States.
Period: Overall Study
Arm/Group | Deoxycholic Acid 2 mg/cm²
Started | 165
Completed | 131 (Completed the last follow-up visit 12 months after last treatment)
Not Completed | 34
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 14
Not completed — Participant Convenience | 10
Not completed — Miscellaneous Reasons | 4

BASELINE CHARACTERISTICS:
Arm/Group | Deoxycholic Acid 2 mg/cm²
Number analyzed (Participants) | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (10.89)
Age, Customized [Number; unit: participants]
  18 - 50 years | 98
  51 - 65 years | 63
  > 65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 37
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 1
  Asian | 7
  Black or African American | 15
  Multiple | 1
  Other | 12
  White | 129
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 30
  Not Hispanic or Latino | 135
Weight [Mean (Standard Deviation); unit: kg] | 80.37 (15.111)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 28.88 (4.311)
Fitzpatrick Skin Type [Number; unit: participants] — Fitzpatrick Skin Type is a numerical classification schema for human skin color and typical response to ultraviolet (UV) light:
  * Type I: Pale white skin, blue/hazel eyes, blond/red hair, always burns, does not tan
  * Type II: Fair skin, blue eyes, burns easily, tans poorly
  * Type III: Darker white skin, tans after initial burn
  * Type IV: Light brown skin, burns minimally, tans easily
  * Type V: Brown skin, rarely burns, tans darkly easily
  * Type VI: Dark brown or black skin, never burns, always tans darkly
  participants
    I - III | 123
    IV - VI | 42
Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) Rating [Number; unit: participants] — CR-SMFRS Ratings:
  * 0 = Absent submental convexity: No localized submental fat evident
  * 1 = Mild submental convexity: Minimal, localized submental fat
  * 2 = Moderate submental convexity: Prominent, localized submental fat
  * 3 = Severe submental convexity: Marked, localized submental fat
  * 4 = Extreme submental convexity
  participants
    2 | 86
    3 | 66
    4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Serious AEs include any event that met one or more of the following criteria: was fatal or life-threatening, required inpatient hospitalization or prolonged a hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or a significant medical hazard.
  The severity of each AE was defined as either:
  Mild: The participant was aware of the sign or symptom, but it was easily tolerated.
  Moderate: The sign or symptom caused discomfort and interfered with usual activity.
  Severe: The sign or symptom was incapacitating, and the participant was unable to engage in usual activity.
  The investigator determined the relationship of each AE to the study drug using the question: "Is there a reasonable possibility that the event may have been caused by treatment with the study drug?"
Time Frame: Up to 12 months after last treatment (maximum of 18 months from first treatment)
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Deoxycholic Acid 2 mg/cm²
Number analyzed (Participants) | 165
participants
  Any adverse event | 160
  Serious adverse event | 7
  Severe adverse event | 11
  Adverse event leading to withdrawal from treatment | 15
  Adverse event leading to study discontinuation | 6
  Adverse event leading to death | 1
  Adverse event related to study drug | 155
  Serious adverse event related to study drug | 0
  Adverse event associated with the treatment area | 158

2. Secondary Outcome: Mean Change From Baseline in Clinician-Reported Submental Fat Rating Scale Scores (CR-SMFRS)
Description: The CR-SMFRS score is based on the investigator's clinical evaluation of the participant, where submental fullness is scored on a 5-point ordinal scale (0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme). A negative change from baseline indicates improvement.
Time Frame: Baseline and months 3, 6, 9, and 12 after last treatment
Population: Treatment effect population (all participants who received at least 1 injection with study drug and had any posttreatment data for treatment effect variables or for the submental skin laxity grade) and with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deoxycholic Acid 2 mg/cm²
Number analyzed (Participants) | 165
units on a scale
  Month 3 after last treatment (n = 144) | -1.3 (0.85)
  Month 6 after last treatment (n = 133) | -1.3 (0.85)
  Month 9 after last treatment (n = 134) | -1.4 (0.81)
  Month 12 after last treatment (n = 131) | -1.4 (0.80)

3. Secondary Outcome: Mean Change From Baseline in Patient-Reported Submental Fat Scale Rating Scale (PR-SMFRS)
Description: The PR-SMFRS is based on the participant's response to the question "How much fat do you have under your chin right now?" and answered on a 5-point ordinal scale (0 = no chin fat at all, 1 = a slight amount of chin fat, 2 = a moderate amount of chin fat, 3 = a large amount of chin fat, and 4 = a very large amount of chin fat). A negative change from baseline indicates improvement.
Time Frame: Baseline and month 3 and month 12 after last treatment
Population: Treatment effect population with available data at baseline (163) and at each time point (indicated by "n")
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deoxycholic Acid 2 mg/cm²
Number analyzed (Participants) | 163
units on a scale
  Month 3 after last treatment (n = 142) | -1.2 (0.90)
  Month 12 after last treatment (n = 127) | -1.3 (0.88)

4. Secondary Outcome: Percentage of Participants Who Achieved a Composite 1-grade Response
Description: A composite 1-grade response is defined as at least a 1-grade improvement from baseline on both the CR-SMFRS and PR-SMFRS.
  The CR-SMFRS score is based on the investigator's clinical evaluation of the participant, where submental fullness is scored on a 5-point ordinal scale (0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme).
  The PR-SMFRS is based on the participant's response to the question "How much fat do you have under your chin right now?" and answered on a 5-point ordinal scale (0 = no chin fat at all, 1 = a slight amount of chin fat, 2 = a moderate amount of chin fat, 3 = a large amount of chin fat, and 4 = a very large amount of chin fat).
Time Frame: Baseline and month 3 and month 12 after last treatment
Population: Treatment effect population with available data at baseline and at each time point (indicated by "n")
Measure: Number; unit: percentage of participants
Arm/Group | Deoxycholic Acid 2 mg/cm²
Number analyzed (Participants) | 163
percentage of participants
  Month 3 after last treatment (n = 142) | 72.5
  Month 12 after last treatment (n = 128) | 75.0

5. Secondary Outcome: Percentage of Participants Who Achieved a Composite 2-grade Response
Description: A composite 2-grade response is defined as at least a 2-grade improvement from baseline on both the CR-SMFRS and PR-SMFRS.
  The CR-SMFRS score is based on the investigator's clinical evaluation of the participant, where submental fullness is scored on a 5-point ordinal scale (0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme).
  The PR-SMFRS is based on the participant's response to the question "How much fat do you have under your chin right now?" and answered on a 5-point ordinal scale (0 = no chin fat at all, 1 = a slight amount of chin fat, 2 = a moderate amount of chin fat, 3 = a large amount of chin fat, and 4 = a very large amount of chin fat).
Time Frame: Baseline and month 3 and month 12 after last treatment
Population: Treatment effect population with available data at baseline and at each time point (indicated by "n")
Measure: Number; unit: percentage of participants
Arm/Group | Deoxycholic Acid 2 mg/cm²
Number analyzed (Participants) | 163
percentage of participants
  Month 3 after last treatment (n = 142) | 14.1
  Month 12 after last treatment (n = 128) | 20.3

6. Secondary Outcome: Mean Change From Baseline in Patient-Reported Submental Fat Impact Scale (PR-SMFIS)
Description: The PR-SMFIS assesses the impact of submental fat on self-perception of 6 emotional and visual characteristics (unhappy, bothered, self-conscious, embarrassed, look older, and look overweight) related to the appearance of submental fullness as evaluated by the participant. Each item is rated on an 11-point numeric scale from 0 to 10. Scores for the 6 items were averaged to generate a PR-SMFIS total scale score ranging from 0 to 10 where 0 is a positive outcome and 10 is a negative outcome. A negative change from baseline indicates improvement.
Time Frame: Baseline and month 3 and month 12 after last treatment
Population: Treatment effect population with available data at baseline and each time point (indicated by "n")
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deoxycholic Acid 2 mg/cm²
Number analyzed (Participants) | 163
units on a scale
  Month 3 after last treatment (n = 145) | -4.3 (2.86)
  Month 12 after last treatment (n = 129) | -4.2 (2.86)

7. Secondary Outcome: Mean Change From Baseline in Subject Self Rating Scale (SSRS)
Description: The SSRS assesses participants' satisfaction with their appearance in association with the face and chin on a 7-point scale from 0 to 6 (0 = extremely dissatisfied, 1 = dissatisfied, 2 = slightly dissatisfied, 3 = neither satisfied nor dissatisfied, 4 = slightly satisfied, 5 = satisfied and 6 = extremely satisfied). A positive change from baseline indicates improvement.
Time Frame: Baseline and month 3 and month 12 after last treatment
Population: Treatment effect population with available data (indicated by "n")
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deoxycholic Acid 2 mg/cm²
Number analyzed (Participants) | 165
units on a scale
  Month 3 after last treatment (n = 144) | 3.6 (1.49)
  Month 12 after last treatment (n = 128) | 3.8 (1.36)

8. Secondary Outcome: Mean Change From Baseline in Self-rating of Attractiveness
Description: Self-rating of Attractiveness assesses aspects of appearance from the participant's perspective with a series of 6 questions: How attractive do you think your overall appearance (chin/neck, eyes, nose, mouth, entire face) is/are?" Each question was answered on a scale from 1 to 9 (1 = not at all attractive, 5 = neither attractive nor unattractive, and 9 = extremely attractive). A positive change from baseline indicates improvement.
Time Frame: Baseline and month 3 and month 12 after last treatment
Population: Treatment effect population with available data at baseline (163), month 3 (144), and month 12 (130)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deoxycholic Acid 2 mg/cm²
Number analyzed (Participants) | 163
units on a scale
  Overall appearance - month 3 after last treatment | 0.8 (1.53)
  Overall appearance - month 12 after last treatment | 1.0 (1.62)
  Chin/neck - month 3 after last treatment | 2.6 (2.35)
  Chin/neck - month 12 after last treatment | 3.1 (2.43)
  Eyes - month 3 after last treatment | 0.4 (1.62)
  Eyes - month 12 after last treatment | 0.6 (1.70)
  Nose - month 3 after last treatment | 0.3 (1.66)
  Nose - month 12 after last treatment | 0.6 (1.97)
  Mouth - month 3 after last treatment | 0.3 (1.45)
  Mouth - month 12 after last treatment | 0.6 (1.44)
  Entire face - month 3 after last treatment | 0.5 (1.27)
  Entire face - month 12 after last treatment | 0.8 (1.28)

9. Secondary Outcome: Response to Subject Global Questions
Description: Participants answered 3 questions on a 7-point scale that ranged from "a great deal worse" to "a great deal better" (questions 1 and 2) or from "extremely dissatisfied" to "extremely satisfied" (question 3).
  Question 1: Since the start of the study, how would you rate the fat under your chin right now?
  Question 2: Since the start of the study, how would you rate the definition between your chin and neck right now?
  Question 3: How satisfied are you with the treatment you received in this study?
Time Frame: Month 3 and month 12 after last treatment
Population: Treatment effect population with available data at each time point
Measure: Number; unit: participants
Arm/Group | Month 3 After Last Treatment | Month 12 After Last Treatment
Number analyzed (Participants) | 145 | 130
participants
  Question 1 - a great deal worse | 0 | 0
  Question 1 - moderately worse | 1 | 1
  Question 1 - a little worse | 0 | 1
  Question 1 - about the same | 6 | 7
  Question 1 - a little better | 22 | 23
  Question 1 - moderately better | 48 | 32
  Question 1 - a great deal better | 68 | 66
  Question 2 - a great deal worse | 0 | 0
  Question 2 - moderately worse | 0 | 1
  Question 2 - a little worse | 0 | 0
  Question 2 - about the same | 5 | 5
  Question 2 - a little better | 27 | 27
  Question 2 - moderately better | 53 | 38
  Question 2 - a great deal better | 60 | 59
  Question 3 - extremely dissatisfied | 1 | 1
  Question 3 - moderately dissatisfied | 0 | 1
  Question 3 - a little dissatisfied | 2 | 2
  Question 3 - neither dissatisfied nor satisfied | 5 | 6
  Question 3 - a little satisfied | 15 | 11
  Question 3 - moderately satisfied | 43 | 30
  Question 3 - extremely satisfied | 79 | 79

10. Secondary Outcome: Percent Change From Baseline in Submental Fat Thickness
Description: Submental fat thickness was measured using calipers.
Time Frame: Baseline and month 3 and month 12 after last treatment
Population: Treatment effect population with available data at baseline (164) and at each time point
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Deoxycholic Acid 2 mg/cm²
Number analyzed (Participants) | 164
percent change
  Month 3 after last treatment (n = 144) | -27.2 (21.82)
  Month 12 after last treatment (n = 131) | -30.9 (20.88)

11. Secondary Outcome: Change From Baseline in Submental Skin Laxity Grade (SMSLG)
Description: SMSLG assessment was based on clinical evaluation and palpation of the submental area. The SMSLG scale incorporates 3 features: skin wrinkling, adherence to underlying neck structures (bone and muscle) and redundancy (horizontal and vertical folds).
  Grade 1 (none): no or minimal superficial wrinkling, skin well apposed to deeper neck structures, no skin redundancy (no skin draping (vertical folds) or skin sagging (horizontal folds));
  Grade 2 (mild): mild superficial wrinkling, skin well apposed to deeper neck structures, minimal skin redundancy (slight skin draping and sagging);
  Grade 3 (moderate): may have mild to moderate superficial wrinkling, skin has mild to moderate separation from deeper neck structures, moderate skin redundancy (moderate skin draping and skin sagging);
  Grade 4 (severe): mild to marked superficial wrinkling, loose skin separated from deeper neck structures, marked skin redundancy (marked skin draping and sagging).
Time Frame: Baseline and month 3 and month 12 after last treatment
Population: Treatment effect population with available data (indicated by "n")
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deoxycholic Acid 2 mg/cm²
Number analyzed (Participants) | 165
units on a scale
  Month 3 after last treatment (n = 144) | -0.3 (0.58)
  Month 12 after last treatment (n = 131) | -0.3 (0.63)

12. Secondary Outcome: Change From Baseline in Line Drawing Assessment
Description: Each participant was given 2 example line drawings representing each of the 5 submental fat grades (0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme) and asked to select the drawing that best represents their current profile. Improvement is any decrease in grade, and worsening is any increase in grade.
Time Frame: Baseline and month 3 after last treatment
Population: Treatment effect population with available data
Measure: Number; unit: participants
Arm/Group | Deoxycholic Acid 2 mg/cm²
Number analyzed (Participants) | 143
participants
  Improved by > 2 | 27
  Improved by 2 | 52
  Improved by 1 | 25
  Unchanged | 31
  Worsened by 1 | 8
  Worsened by 2 | 0
  Worsened by > 2 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months after last treatment (maximum of 18 months from first treatment)
Arm/Group | Deoxycholic Acid 2 mg/cm²
Serious Adverse Events (participants affected / at risk) | 7/165
Other Adverse Events (participants affected / at risk) | 160/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deoxycholic Acid 2 mg/cm² (N=165)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardiac death (General disorders) | 1
Diverticulitis (Infections and infestations) | 1
Anxiety (Psychiatric disorders) | 1
Cervical polyp (Reproductive system and breast disorders) | 1
Stent placement (Surgical and medical procedures) | 1
Arteriosclerosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deoxycholic Acid 2 mg/cm² (N=165)
Injection site hematoma (General disorders) | 121
Injection site anesthesia (General disorders) | 116
Injection site pain (General disorders) | 113
Injection site edema (General disorders) | 111
Injection site erythema (General disorders) | 83
Injection site induration (General disorders) | 61
Injection site swelling (General disorders) | 49
Injection site pruritus (General disorders) | 36
Injection site nodule (General disorders) | 32
Injection site paresthesia (General disorders) | 31
Headache (Nervous system disorders) | 15
Blood triglycerides increased (Investigations) | 12
Blood glucose increased (Investigations) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical study agreement requires that the investigator or institution obtain written consent from Kythera Biopharmaceuticals, Inc. prior to presenting and/or publishing results of this study.